CLINICAL TRIAL: NCT06515639
Title: Classic vs. High-Fat Intermittent Fasting: Impacts on Body Composition, Eating Behavior, and Diet Satisfaction
Brief Title: Classic vs. High-Fat Intermittent Fasting Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Emre Batuhan Kenger, Assistant Prof., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IFLOWCARB
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Obesity
Keywords: Intermittent fasting diet; body composition; eating behavior; diet satisfaction
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic IF diet (Experimental): The 16:8 intermittent fasting model, 45-60% carbohydrates, 10-15% protein, and 25-30% fat dietary model applied.
  Interventions: Other: Diet therapy for Classic IF diet group
- Low carb-High fat IF diet (Experimental): The 16:8 intermittent fasting model, 10-30% carbohydrates and 50-65% fat dietary model applied.
  Interventions: Other: Diet therapy for low carb-High fat IF diet group

INTERVENTIONS:
Other: Diet therapy for Classic IF diet group — The 16:8 intermittent fasting model was applied for six weeks. Time restrictions were tailored to fit the participants' lifestyles, with feeding times set between 10:00-12:00 and 18:00-20:00 for all participants. The classic intermittent fasting diet was planned with a macronutrient distribution of 45-60% carbohydrates, 10-15% protein, and 25-30% fat. Additionally, total energy intake was reduced by 500-750 kcal.
  Arms: Classic IF diet
Other: Diet therapy for low carb-High fat IF diet group — The 16:8 intermittent fasting model was applied for six weeks. Time restrictions were tailored to fit the participants' lifestyles, with feeding times set between 10:00-12:00 and 18:00-20:00 for all participants.The low carb-high fat intermittent fasting diet included 10-30% carbohydrates and 50-65% fat.Additionally, total energy intake was reduced by 500-750 kcal.
  Arms: Low carb-High fat IF diet

SUMMARY:
Poor eating habits contribute to weight gain and obesity, leading to numerous metabolic issues such as diabetes and cardiovascular diseases. The treatment of obesity involves lifestyle interventions that include dietary and nutritional modifications, physical activity, and behavioral therapy. Literature supports both carbohydrate and fat restriction in the treatment of obesity. In low-carbohydrate diets, less than 40% of energy is sourced from carbohydrates.Besides the dietary model, individual eating behavior can also influence the diet's outcomes. There is a significant relationship between eating behavior and food choices. Given that food choices can impact diet satisfaction, evaluating eating behavior is important when assessing dietary compliance.The literature includes studies demonstrating the effects of a classic intermittent fasting diet. However, no studies have compared the potential effects of intermittent fasting models based on the macronutrient distribution within their content. Therefore, this study aims to evaluate the effects of high-fat, low-carbohydrate intermittent fasting versus classical intermittent fasting on body composition, eating behavior, and diet satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* no chronic disease
* female
* volunteering

Exclusion Criteria:

* hypoglycemia
* eating disorders
* pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Body composition | six weeks
  measurements of total body weight
Body composition | six weeks
  measurements of body mass index (BMI)
Body composition | six weeks
  measurements of fat mass
Body composition | six weeks
  measurements of muscle mass
Body composition | six weeks
  measurements of fat percentage
diet satisfaction | six weeks
  A number of questions are necessary for clinicians to evaluate their patients' or clients' diet satisfaction, as well as their compliance with the diet, based on their responses. The Diet Satisfaction Scale is designed to assess satisfaction with various aspects of any diet, such as hunger levels, desire to eat, food preparation, enjoyment, ease of adherence at home and away, food variety, budget compatibility, contribution to physical health, and sustainability. The scale was developed by Jospe et al, and its Turkish validity and reliability were established by Eskici and Yilmaz. It consists of 9 items with 5-point Likert-type response options ranging from 1 (strongly disagree) to 5 (strongly agree). Notably, the first item is reverse-scored (1=5, 2=4, 3=3, 4=2, and 5=1).
behavioral and cognitive components of eating | six weeks
  The Three-Factor Eating Scale, used to measure the behavioral and cognitive components of eating, was developed by Cappelleri and colleagues. Its validity and reliability in Turkish were established by Karakus et al. The questionnaire comprises three factors: Uncontrolled Eating (UE), Cognitive Restraint (CR), and Emotional Eating (EE). Uncontrolled Eating (UE) refers to losing control over eating due to hunger or external stimuli and includes 9 items, with scores ranging from 9 to 36. Cognitive Restraint (CR) refers to the conscious restriction of food intake to control body shape and weight, encompassing 6 items, with scores ranging from 6 to 24. Emotional Eating (EE) examines overeating in response to negative emotional states such as anger, sadness, or stress, and includes 6 items, with scores ranging from 6 to 24. A higher score in any sub-factor indicates a greater dominance of the corresponding eating behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Gebze Municipality Family Counseling Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared if requested by the authors.

REFERENCES:
- [Background] Konttinen H. Emotional eating and obesity in adults: the role of depression, sleep and genes. Proc Nutr Soc. 2020 Aug;79(3):283-289. doi: 10.1017/S0029665120000166. Epub 2020 Mar 26. PMID 32213213
- [Background] Wadden TA, Tronieri JS, Butryn ML. Lifestyle modification approaches for the treatment of obesity in adults. Am Psychol. 2020 Feb-Mar;75(2):235-251. doi: 10.1037/amp0000517. PMID 32052997
- [Background] Willems AEM, Sura-de Jong M, van Beek AP, Nederhof E, van Dijk G. Effects of macronutrient intake in obesity: a meta-analysis of low-carbohydrate and low-fat diets on markers of the metabolic syndrome. Nutr Rev. 2021 Mar 9;79(4):429-444. doi: 10.1093/nutrit/nuaa044. PMID 32885229
- [Background] Flaskerud JH. Mood and food. Issues Ment Health Nurs. 2015 Apr;36(4):307-10. doi: 10.3109/01612840.2014.962677. No abstract available. PMID 25988966
- [Background] Welton S, Minty R, O'Driscoll T, Willms H, Poirier D, Madden S, Kelly L. Intermittent fasting and weight loss: Systematic review. Can Fam Physician. 2020 Feb;66(2):117-125. PMID 32060194
- [Background] Cappelleri JC, Bushmakin AG, Gerber RA, Leidy NK, Sexton CC, Lowe MR, Karlsson J. Psychometric analysis of the Three-Factor Eating Questionnaire-R21: results from a large diverse sample of obese and non-obese participants. Int J Obes (Lond). 2009 Jun;33(6):611-20. doi: 10.1038/ijo.2009.74. Epub 2009 Apr 28. PMID 19399021
- [Background] Karakuş SS, Yıldırım H, Büyüköztürk Ş. Adaptation of the Three-Factor Eating Questionnaire into Turkish: A validity and reliability study. Prev Med Bull 2016;15, 229-237.
- [Background] Jospe MR, Haszard JJ, Taylor RW, Freedhoff Y. A tool for assessing the satisfaction of a diet: Development and preliminary validation of the Diet Satisfaction Score. Nutr Diet. 2020 Apr;77(2):268-273. doi: 10.1111/1747-0080.12591. Epub 2019 Nov 3. PMID 31680438
- [Background] Eskici G, Yılmaz SK. Validity and reliability study of the Turkish form of the Diet Satisfaction Scale. Ankara Sağlık Bilim Derg 2021; 10, 35-45.